CLINICAL TRIAL: NCT03023085
Title: A Pilot Evaluation of BLI4700 Bowel Preparation in Adult Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLI4700-201
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BLI4700 (Experimental): BLI4700 Bowel Preparation
  Interventions: Drug: BLI4700

INTERVENTIONS:
Drug: BLI4700 — BLI4700 bowel preparation

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of BLI4700 as a bowel preparation prior to colonoscopy in adult patients.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication.
2. Have previously had a colonoscopy performed
3. At least 18 years of age
4. Subjects must be scheduled for a morning colonoscopy (prior to 12:00PM)
5. If female, and of child-bearing potential, is using an acceptable form of birth control.
6. Negative urine pregnancy test at screening, if applicable
7. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Key Exclusion Criteria:

1. Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
2. Subjects who had previous significant gastrointestinal surgeries.
3. Subjects with uncontrolled pre-existing electrolyte abnormalities, or those with clinically significant electrolyte abnormalities based on Visit 1 laboratory results.
4. Subjects with a prior history of renal, liver or cardiac insufficiency
5. Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
6. Subjects undergoing colonoscopy for foreign body removal and/or decompression.
7. Subjects who are pregnant or lactating, or intending to become pregnant during the study.
8. Subjects of childbearing potential who refuse a pregnancy test.
9. Subjects allergic to any preparation components.
10. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
11. Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (1):
- Braintree Research Site 1, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BLI4700 (Study Formulation 1); BLI4700 (Study Formulation 2); BLI4700 (Study Formulation 3); BLI4700 (Study Formulation 4): BLI4700 Bowel Preparation
  BLI4700: BLI4700 tablet bowel preparation
Period: Overall Study
Arm/Group | BLI4700 (Study Formulation 1) | BLI4700 (Study Formulation 2) | BLI4700 (Study Formulation 3) | BLI4700 (Study Formulation 4)
Started | 40 | 37 | 17 | 20
Completed | 38 | 26 | 17 | 19
Not Completed | 2 | 11 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI4700 (Study Formulation 1) | BLI4700 (Study Formulation 2) | BLI4700 (Study Formulation 3) | BLI4700 (Study Formulation 4) | Total
Number analyzed (Participants) | 40 | 37 | 17 | 20 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (11.9) | 59.8 (9.8) | 58.3 (9.1) | 56.6 (10.6) | 58.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 12 | 12 | 67
  Male | 21 | 13 | 5 | 8 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 4 | 0 | 3 | 18
  Not Hispanic or Latino | 29 | 33 | 17 | 17 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 11 | 3 | 2 | 18
  White | 37 | 25 | 14 | 18 | 94
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 37 | 17 | 20 | 114

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects With Successful Bowel Cleansing
Description: % of subjects with successful bowel preparation rated by blinded colonoscopist on a 4 point scale (1=poor, 2=fair, 3=good, 4 = excellent)
Time Frame: Day of colonoscopy
Population: Efficacy population - all patients that took any portion of the preparation and did not discontinue from the study for a reason other than safety or efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | BLI4700 (Study Formulation 1) | BLI4700 (Study Formulation 2) | BLI4700 (Study Formulation 3) | BLI4700 (Study Formulation 4)
Number analyzed (Participants) | 40 | 37 | 17 | 20
Participants | 35 | 36 | 16 | 19

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | BLI4700 (Study Formulation 1) | BLI4700 (Study Formulation 2) | BLI4700 (Study Formulation 3) | BLI4700 (Study Formulation 4)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/37 | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/37 | 0/17 | 1/20
Other Adverse Events (participants affected / at risk) | 30/40 | 24/37 | 12/17 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI4700 (Study Formulation 1) (N=40) | BLI4700 (Study Formulation 2) (N=37) | BLI4700 (Study Formulation 3) (N=17) | BLI4700 (Study Formulation 4) (N=20)
Syncope (Nervous system disorders) | NA | NA | NA | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BLI4700 (Study Formulation 1) (N=40) | BLI4700 (Study Formulation 2) (N=37) | BLI4700 (Study Formulation 3) (N=17) | BLI4700 (Study Formulation 4) (N=20)
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 19 | 18 | 9 | 13 — Study subjects were queried by research staff for this expected preparation symptom.
Vomiting (Gastrointestinal disorders) | 10 | 6 | 3 | 4 — Study subjects were queried by research staff for this expected preparation symptom.
Abdominal Pain (Gastrointestinal disorders) | 9 | 12 | 3 | 4 — Study subjects were queried by research staff for this expected preparation symptom.
Abdominal Distension (Gastrointestinal disorders) | 11 | 18 | 6 | 8 — Study subjects were queried by research staff for this expected preparation symptom.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT03023085/Prot_SAP_000.pdf